CLINICAL TRIAL: NCT00003724
Title: Phase III Randomized Prospective Trial of Open Versus Minimally Invasive, Video-Assisted Resection of Pulmonary Metastases
Brief Title: Conventional or Video-Assisted Surgery in Treating Patients With Lung Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39804; U10CA031946 (NIH); CLB-39804; CDR0000066833 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Cancer
Keywords: lung metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery (Experimental): Patients undergo open resection (thoracotomy, median sternotomy, or bilateral sternothoracotomy).
  Patients with isolated recurrence in the chest should have the recurrence(s) resected if feasible. The original resection approach (open versus VATS) should be the preferred method for the second resection, but is not required.
  Quality of life is assessed prior to randomization and then at 30 days, 3 months, and 6 months. Patients are followed every 3 months for 1 year and then every 6 months thereafter.
  Interventions: Procedure: surgical procedure
- video-assisted surgery (Experimental): After spiral CT showing pulmonary nodules are amenable to video-assisted thoracic surgery (VATS) resection with curative intent, patients undergo minimally-invasive video-assisted resection.
  Patients with isolated recurrence in the chest should have the recurrence(s) resected if feasible. The original resection approach (open versus VATS) should be the preferred method for the second resection, but is not required.
  Quality of life is assessed prior to randomization and then at 30 days, 3 months, and 6 months. Patients are followed every 3 months for 1 year and then every 6 months thereafter.
  Interventions: Procedure: surgical procedure

INTERVENTIONS:
Procedure: surgical procedure

SUMMARY:
RATIONALE: Video-assisted surgery may have fewer side effects than conventional surgery in patients with lung metastases. It is not yet known whether conventional surgery or video-assisted surgery is more effective in treating lung metastases.

PURPOSE: Randomized phase III trial to compare the effectiveness of conventional surgery with that of video-assisted surgery in treating patients who have lung metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival and failure free survival of patients with isolated pulmonary metastases treated with minimally invasive (video assisted) resection or open resection. II. Compare patterns of recurrence in these patients after these treatments, and determine what factors are predictive of recurrence. III. Describe and compare the complications and morbidity associated with minimally-invasive and open approaches to metastasectomy in these patients. IV. Test whether the patients undergoing video-assisted thoracic surgery will have a significantly better quality of life over a six month period than those undergoing an open resection.

OUTLINE: This is a randomized study. Patients are stratified according to histology (sarcoma vs epithelial vs germ cell vs melanoma) and disease laterality. After spiral CT showing pulmonary nodules are amenable to video-assisted thoracic surgery (VATS) resection with curative intent, patients are randomized to undergo either open resection (thoracotomy, median sternotomy, or bilateral sternothoracotomy) (arm I) or minimally-invasive video-assisted resection (arm II). Patients with isolated recurrence in the chest should have the recurrence(s) resected if feasible. The original resection approach (open versus VATS) should be the preferred method for the second resection, but is not required. Quality of life is assessed prior to randomization and then at 30 days, 3 months, and 6 months. Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: There will be 530 patients accrued into this study in approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed pulmonary metastases (unilateral or bilateral) identified by spiral CT scan No primary lung cancer Documented previous cancer with no history of prior metastasectomy Primary tumor must be definitively controlled No evidence of primary tumor recurrence, either locally or systemically No extrapulmonary metastatic disease or evidence of mediastinal lymph node involvement Lymph nodes greater than 1.0 cm on CT scan must be proven to be benign by tissue biopsy (mediastinoscopy) All lesions must be amenable to minimally invasive resection Must be amenable to video-assisted thoracic surgery with curative intent (complete removal of all documented lesions) No greater than 4 lesions

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Pulmonary: See Disease Characteristics

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 1999-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 5 years

SECONDARY OUTCOMES:
recurrence free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R. Sonett, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (45):
- United States (45):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - University of Missouri, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia